CLINICAL TRIAL: NCT01072123
Title: Innovative Asthma Education Using a Unique Blend of Child Life Services and an Asthma-based Computer Game in the Pediatric Emergency Room
Brief Title: Asthma Education Using Child Life Services and an Asthma-based Computer Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 08313
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Quest for the Code — interactive asthma-based computer program

SUMMARY:
This is a single center pilot study designed to evaluate the effectiveness of an asthma education program in the pediatric emergency department. Asthma has reached epidemic proportions. Nine million American children are affected in the United States alone. This problem has increased 75% from 1980 to 1994, with a staggering 160% increase seen in children less than five years old.1 The American Lung Association has targeted this overwhelming problem on both national and local levels. Asthma impacts American communities who differ geographically, culturally, ethnically and by lifestyle, and as a result will present with different obstacles.

The primary objectives are: to determine whether this educational intervention (through interactions with a child life specialist and using the asthma based computer game) in the pediatric ED can influence children's [and care givers'] knowledge and understanding of the disease process and treatment, and to improve asthma self-management and decrease morbidity by decreasing ED use and hospitalization.

A secondary objective is to introduce the Child Life Specialist as an effective asthma educator and further strengthen the health care team.

The target population will be recruited from the pediatric emergency department. We anticipate this study to recruit over a one year period and have a one year follow up with an anticipated enrollment of 64 children and families. There will be three Child Life Specialist involved in this program.

After consent has been obtained, the child and parent will complete questionnaires (focusing on asthma knowledge, quality of life, and perception of asthma) and then a laptop will be provided to access the asthma based computer game.

During the child's ED visit the Child Life Specialist will have opportunities to open communication to address barriers or concerns, and reinforce material provided by the game. Through these interactions, the importance of communication between the child, parent and healthcare provider is highlighted.

The family will be given information to access the computer game via the internet. Follow up phone calls or e-mails will occur at 6 months, 9 months, and 12 months which will entail completing questionnaires. The questionnaires uses validated questions along with questions from the material covered through this asthma education study.

ELIGIBILITY:
Inclusion Criteria:

* Age between six to eighteen years old
* Diagnosis of asthma

Exclusion Criteria:

* Refused to participate in the study
* Unable to understand or respond to questions
* If participants are not English speaking

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine whether an educational intervention in the pediatric ED or during hospitalization can influence children's [and care givers'] knowledge and understanding of the disease process and treatment. | 1 year
To improve communication, asthma self-management and decrease morbidity by decreasing ED use and hospitalization | 1 year

SECONDARY OUTCOMES:
To introduce the Child Life Specialist as an effective asthma educator and further strengthen the health care team | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cataletto, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Gupta RS, Zhang X, Sharp LK, Shannon JJ, Weiss KB. Geographic variability in childhood asthma prevalence in Chicago. J Allergy Clin Immunol. 2008 Mar;121(3):639-645.e1. doi: 10.1016/j.jaci.2007.11.036. Epub 2008 Feb 4. PMID 18243285
- [Background] Smeeton NC, Rona RJ, Gregory J, White P, Morgan M. Parental attitudes towards the management of asthma in ethnic minorities. Arch Dis Child. 2007 Dec;92(12):1082-7. doi: 10.1136/adc.2006.112037. Epub 2007 Feb 6. PMID 17284478
- [Background] Zayas LE, McLean D. Asthma patient education opportunities in predominantly minority urban communities. Health Educ Res. 2007 Dec;22(6):757-69. doi: 10.1093/her/cyl070. Epub 2006 Aug 8. PMID 16896054
- [Background] Wakefield M, Staugas R, Ruffin R, Campbell D, Beilby J, McCaul K. Risk factors for repeat attendance at hospital emergency departments among adults and children with asthma. Aust N Z J Med. 1997 Jun;27(3):277-84. doi: 10.1111/j.1445-5994.1997.tb01979.x. PMID 9227811
- [Background] Wasilewski Y, Clark NM, Evans D, Levison MJ, Levin B, Mellins RB. Factors associated with emergency department visits by children with asthma: implications for health education. Am J Public Health. 1996 Oct;86(10):1410-5. doi: 10.2105/ajph.86.10.1410. PMID 8876510
- [Background] Franks TJ, Burton DL, Simpson MD. Patient medication knowledge and adherence to asthma pharmacotherapy: a pilot study in rural Australia. Ther Clin Risk Manag. 2005 Mar;1(1):33-8. doi: 10.2147/tcrm.1.1.33.53598. PMID 18360541
- [Background] Flores G, Abreu M, Tomany-Korman S, Meurer J. Keeping children with asthma out of hospitals: parents' and physicians' perspectives on how pediatric asthma hospitalizations can be prevented. Pediatrics. 2005 Oct;116(4):957-65. doi: 10.1542/peds.2005-0712. PMID 16199708
- [Background] Cagan ER, Hubinsky T, Goodman A, Deitcher D, Cohen NL. Partnering with communities to improve health: the New York City Turning Point experience. J Urban Health. 2001 Mar;78(1):176-80. doi: 10.1093/jurban/78.1.176. PMID 11368196
- [Background] Lara M, Rosenbaum S, Rachelefsky G, Nicholas W, Morton SC, Emont S, Branch M, Genovese B, Vaiana ME, Smith V, Wheeler L, Platts-Mills T, Clark N, Lurie N, Weiss KB. Improving childhood asthma outcomes in the United States: a blueprint for policy action. Pediatrics. 2002 May;109(5):919-30. doi: 10.1542/peds.109.5.919. PMID 11986457
- [Background] Persky V, Coover L, Hernandez E, Contreras A, Slezak J, Piorkowski J, Curtis L, Turyk M, Ramakrishnan V, Scheff P. Chicago community-based asthma intervention trial: feasibility of delivering peer education in an inner-city population. Chest. 1999 Oct;116(4 Suppl 1):216S-223S. doi: 10.1378/chest.116.suppl_2.216s. PMID 10532497
- [Background] Krishna S, Francisco BD, Balas EA, Konig P, Graff GR, Madsen RW; Randomized trial. Internet-enabled interactive multimedia asthma education program: a randomized trial. Pediatrics. 2003 Mar;111(3):503-10. doi: 10.1542/peds.111.3.503. PMID 12612228
- See also: game — http://www.starlight.org